CLINICAL TRIAL: NCT07234305
Title: Shock Wave Therapy Versus Conventional Physical Therapy for Partial- Thickness Forearm Burn Scars
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MTI University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Ahmed Abd El hady El Fahl,ph.d, Assisstant professor, MTI University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00014233-52
Record Dates: First submitted 2025-11-14; First posted 2025-11-18 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Burn Scar; Burns
MeSH Terms: conditions — Burns

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant
Masking Description: single blinded
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Shock wave (Experimental): The treatment regimen included 2000 shocks directed to the 10 cm2 scar tissue itself, 1000 shocks to the surrounding soft tissue to promote healing. Pneumatic extracorporeal shock wave therapy (ESWT) will administered using the EME Srl device (Via Degli Abeti, Pesaro- Italy) over a series of sessions
  Interventions: Other: Shock wave
- Traditional Physical Therapy (Experimental): This included five minutes of passive stretching for the wrist flexors, with therapist assistance, followed by five minutes of active stretching, encouraging patients to engage in movements independently to enhance flexibility and alleviate stiffness. To rebuild strength and functionality in the forearm and hand, the regimen incorporated progressive resistance exercises such as wrist flexion and extension, performed for 20 repetitions per set, two sets per session, three times weekly, using light weights (Vinyl Dumbbell Set, Soft Grips - 2kg, progressing to 3kg, made in China). Grip strengthening exercises were also included, utilizing a guitar finger exercise grip (made in China), with 30 repetitions per set, two sets per day, three times a week.
  Interventions: Other: Traditional Physical Therapy

INTERVENTIONS:
Other: Shock wave — The treatment regimen will include2000 shocks directed to the 10 cm2 scar tissue itself, 1000 shocks to the surrounding soft tissue to promote healing. Pneumatic extracorporeal shock wave therapy (ESWT) will administered using the EME Srl device (Via Degli Abeti, Pesaro- Italy) over a series of sessions. Patients received two sessions each week for 8 successive weeks
  Arms: Shock wave
Other: Traditional Physical Therapy — This included five minutes of passive stretching for the wrist flexors, with therapist assistance, followed by five minutes of active stretching, encouraging patients to engage in movements independently to enhance flexibility and alleviate stiffness. To rebuild strength and functionality in the forearm and hand, the regimen incorporated progressive resistance exercises such as wrist flexion and extension, performed for 20 repetitions per set, two sets per session, three times weekly, using light weights (Vinyl Dumbbell Set, Soft Grips - 2kg, progressing to 3kg, made in China). Grip strengthening exercises were also included, utilizing a guitar finger exercise grip (made in China), with 30 repetitions per set, two sets per day, three times a week.
  Arms: Traditional Physical Therapy

SUMMARY:
Burn injuries can lead to significant physical and psychological challenges, particularly when they result in scarring. Burn scars can lead to a variety of complications that significantly impact a patient's quality of life1.

Physical complications often include restricted range of motion and contractures, which can hinder mobility and daily activities, especially if the scars are located near joints2. Additionally, psychosocial effects such as anxiety, depression, and social withdrawal may arise due to the visible nature of scars and the stigma associated with them3.

Functional complications can also manifest, affecting the skin's ability to regulate temperature and moisture, increasing susceptibility to infections, and causing discomfort or pain 4. In some cases, burn scars may develop into hypertrophic scars or keloids, leading to further aesthetic concerns and potential need for medical interventions5.

Among the various types of burns, partial thickness burns are particularly concerning due to their potential for hypertrophic scarring and functional limitations6. Effective treatment strategies are essential to manage these scars, promote healing, and improve the quality of life for affected individuals7.

DETAILED DESCRIPTION:
Ultrasonography has emerged as a valuable tool in the assessment and monitoring of scar tissue characteristics, allowing for non-invasive evaluation of tissue composition, vascularity, and changes over time. This imaging modality provides critical insights into the healing process, facilitating more informed therapeutic decisions8.

Shock wave therapy has gained attention in recent years as a novel treatment option for scar management. It utilizes acoustic waves to stimulate tissue regeneration, enhance blood flow, and promote collagen remodeling, potentially leading to improved scar quality9.

In contrast, traditional physical therapy remains a cornerstone of rehabilitation post-burn, focusing on restoring function, reducing pain, and improving mobility through various modalities, including stretching, strengthening, and manual therapy techniques 10.

This research addresses the limited exploration of the comparative effectiveness of shock wave therapy versus traditional physical therapy in treating partial thickness burn scars on the forearm. By utilizing a prospective randomized clinical trial design, the study aims to provide substantial evidence regarding the efficacy of these two treatment modalities. The primary focus is to evaluate the impact of both therapies on scar characteristics, specifically examining changes in echogenicity, vascularity, and overall morphology through ultrasonography before and after treatment. Additionally, the study seeks to compare patient-reported outcomes related to scar appearance, pain, and functional abilities between the two groups, ultimately contributing to the development of improved treatment protocols for burn scars.

ELIGIBILITY:
Inclusion Criteria:

* adults diagnosed with partial thickness burns on the forearm,
* scars that had been present for a minimum of six months,
* participants capable of providing informed consent

Exclusion Criteria:

* hypersensitivity to shock wave therapy,
* active infections at the burn site,
* neurological disorders that could impact sensation,
* any contraindications that would prevent the use of ultrasonography.

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2025-10-01 (Actual); Primary Completion 2026-02-01 (Actual); Study Completion 2026-02-04 (Actual)

PRIMARY OUTCOMES:
Ultrasonography Assessment | at baseline , at 8 weeks and 8 weeks follow up
  High-resolution ultrasound was performed using the GE Logiq P6 Pro (GE Healthcare, Solingen, Germany) machine, to measure scars during the pre-treatment, post-treatment, and follow-up periods. Scar thickness is determined at the thickest point of irregular scars
The Vancouver Scar Scale | at baseline, at 8 weeks and 8 weeks follow up
  The total score can range from 0 to 13, where a score of zero indicates normal skin and a score of 13 reflects the most worse scar tissue. In this study, the VSS was utilized to assess forearm scars in participants at baseline before any interventions, again after 8 weeks of treatment, and finally 8 weeks post-intervention to monitor changes over time12.

SECONDARY OUTCOMES:
The Burn Specific Health Scale-Brief (BSHS-B) | at baseline , at 8 weeks and 8 weeks follow up
  The questionnaire is divided into nine sub-domains, which cover areas such as emotional well-being, basic abilities, employment, social interactions, heat sensitivity, sexual health, treatment processes, self-image, and upper limb functionality. Respondents use a 5-point Likert scale to indicate the level of difficulty or impact related to their burn experiences. The BSHS-B effectively captures the complexities of recovery and distress following burns. BSHS-B was utilized to assess forearm scars in participants at baseline before any interventions, again after 8 weeks of treatment, and finally 8 weeks' post-intervention to monitor changes over time13.

CONTACTS AND LOCATIONS:
Locations (1):
- faculty of physical therapy ,Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No